CLINICAL TRIAL: NCT05495451
Title: Feasibility and Impact of an Intensive Team-based Intervention on Type 2 Diabetes Reversal
Acronym: DIABEPIC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Louis Bherer, Director of Centre EPIC research lab, Montreal Heart Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICM 2022-3018
Record Dates: First submitted 2022-03-14; First posted 2022-08-10 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Type 2 Diabetes
Keywords: Mediterranean Diet, Intermittent Fasting, Training, Lifestyle Changes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: 36 participants will be taught to follow the Mediterranean diet (40% carbohydrates) and training 3 times a week (HIIT and weight training) for 3 months. At 3 months, there will be a randomization: 12 participants will continue the same interventions while 24 will add Intermittent Fasting Intervention for 3 months.
Who Masked: Outcomes Assessor
Masking Description: The randomisation will be effectuated with the participant number only for the Intermittent Fasting Intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean diet and Personalized training (Experimental): 36 participants will participate to the following lifestyle changes for 6 months:
  Behavioral: Lifestyle changes Nutritional advice to progressively integrate a moderate-carbohydrate Mediterranean diet.
  Personalized exercise prescription and training (3 times per week)
  Personalized education and motivational interviewing
  Interventions: Behavioral: Moderate-carbohydrate Mediterranean diet, Personalized exercice prescription and training, Intermittent fasting
- Intermittent Fasting Intervention (Active Comparator): Between 3 and 6 months, 24 participants (on a total of 36) will progressively integrate intermittent fasting 16:8 (5 times/week for 12 weeks) and 20:4 (2 times/week for 4 weeks)
  Interventions: Behavioral: Moderate-carbohydrate Mediterranean diet, Personalized exercice prescription and training, Intermittent fasting

INTERVENTIONS:
Behavioral: Moderate-carbohydrate Mediterranean diet, Personalized exercice prescription and training, Intermittent fasting — Multidisciplinary program will provide the teaching and supervision necessary to integrate the new knowledge and commitment to these lifestyle changes.

SUMMARY:
To evaluate the feasibility of a 6-month multidisciplinary program to reverse type 2 diabetes using the Mediterranean diet, intermittent fasting and exercise.

DETAILED DESCRIPTION:
The morbidities associated with type 2 diabetes (Db2) are major, including cardiovascular and renal complications, but also cognitive impairment. Providing interventions targeting Db2 reversal has shown great potential to improve healthy aging.

A Db2 reversal clinic has been established at the Montreal Heart Institute's ÉPIC Center, with an approach based on the Mediterranean diet and exercise. First-year results showed a 0.6% decrease in Hb1Ac and an average weight loss at 3 months of 4.5 kg in diabetic patients. This improvement was maintained at 6 and 12 months. Although these results are encouraging, the literature in Db2 remission shows that a weight loss of 10 kg is the ideal goal.

Therefore, to offer the possibility of further metabolic improvement at 6 months, three interventions are proposed as additions to the current program: targeting ultra-processed food reduction, motivational coaching and intermittent fasting. The main objective of our pilot study is to determine the feasibility of this improved program in type 2 diabetic patients, aged 18 to 80 years.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Ability to give written consent, to use a smartphone application or complete an adherence/compliance diary, and use a blood glucose and blood pressure machine at home.

Exclusion Criteria:

* All types of diabetes other than type 2
* Taking the following glucose-lowering agents: insulin, sulfonylureas
* BMI < 18,5 kg/m2
* Unintentional weight loss of more than 10 kg in the past year
* Moderate to severe retinopathy
* Pregnant or nursing woman
* Severe organ failure
* Pathologies predisposing to gastrointestinal bleeding, untreated
* Recent cholecystitis (3 months)
* Antibiotic use in the past 3 months, or untreated active infection
* Known impaired nutrient absorption
* Uninvestigated new anemia or Hb < 110 g/100 mL
* Currently following an intermittent or prolonged fasting protocol
* Currently following a specific diet (vegan, celiac/gluten free, ketogenic)
* Active diagnoses of psychiatric or neurological illness not controlled for at least 6 months
* Taking, stopping or adjusting a medication in the last 3 months resulting in an active weight change.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-01-21 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-05-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of an intensive multidisciplinary program based on lifestyle changes in patients diagnosed with type 2 diabetes. | at 3 months after the start of the intervention
  Total recruitment, recruitment rate, compliance and completion rate at 3 months after the start of the intervention
Feasibility of an intensive multidisciplinary program based on lifestyle changes in patients diagnosed with type 2 diabetes. | at 6 months after the start of the intervention
  Total recruitment, recruitment rate, compliance and completion rate at 6 months after the start of the intervention

SECONDARY OUTCOMES:
Proportion of diabetic participants in complete remission of diabetes. | at 3 and 6 months of the start of the intervention
  Remission of diabetes will be defined by the following 3 criteria:
  1. An HbA1c < 6,5% at 3 months of intervention (Metabolic criteria)
  2. Which is maintained at 6 months (Duration criteria)
  3. Without the use of glucose-lowering agents (Pharmacological criteria)
  Proportion of prediabetic patients that reach an Hb1Ac < 6,5% at 6 months of intervention will also be studied
Evolution of the HOMA-IR between the start of the program, the middle of the intervention (3 months) and the end of the intervention (6 months). | at 3 and 6 months of the start of the intervention
  HOMA-IR is a marker of insulin resistance

CONTACTS AND LOCATIONS:
Locations (1):
- EPIC Center of the Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
If the sponsor accepts, we would agree with making individual date available to other researchers
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: One year after completion of the study
Access Criteria: Upon request to the principal investigator

REFERENCES:
- See also: Lean ME, Leslie WS, Barnes AC, Brosnahan N, Thom G, Mccombie L, et al.. Primary care-led weight management for remission of type 2 diabetes (DiRECT): an open-label, cluster-randomised trial. The Lancet 2018;391:541-51. doi:10.1016/s0140-6736(17)33102-1. — http://pubmed.ncbi.nlm.nih.gov/29221645
- See also: Taylor R, Al-Mrabeh A, Sattar N. Understanding the mechanisms of reversal of type 2 diabetes. Lancet Diabetes Endocrinol. 2019 Sep;7(9):726-736. — http://pubmed.ncbi.nlm.nih.gov/31097391
- See also: Zhyzhneuskaya SV, Al-Mrabeh A, Peters C et al. Time Course of Normalization of Functional β-Cell Capacity in the Diabetes Remission Clinical Trial After Weight Loss in Type 2 Diabetes. Diabetes Care 2020;43:813-2 — http://pubmed.ncbi.nlm.nih.gov/32060017
- See also: Kemps H, Kränkel N, Dörr M et al.. Exercise training for patients with type 2 diabetes and cardiovascular disease: What to pursue and how to do it. A Position Paper of the European Association of Preventive Cardiology — http://pubmed.ncbi.nlm.nih.gov/30642190
- See also: de Cabo R, Mattson MP. Effects of Intermittent Fasting on Health, Aging, and Disease. N Engl J Med. 2019 Dec 26;381(26):2541-2551 — http://pubmed.ncbi.nlm.nih.gov/31881139